CLINICAL TRIAL: NCT05780931
Title: Development of New Approaches to Rehabilitating Vision Loss in Veterans With Age-Related Macular Degeneration
Brief Title: Rehabilitating Vision Loss in Veterans With Age-Related Macular Degeneration
Acronym: AMD
Status: Not yet recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Augusta University (Other)
Responsible Party: Sponsor
Other Study IDs: C4099-P; I21RX004099-01A1 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: Maculopathy; Macular dystrophy; Drusen; wet AMD; dry AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: This is the group of study subjects which will undergo study-related rehabilitation procedures.
  Interventions: Behavioral: Study-specific rehabilitation (SSR) procedures
- Control Group: This is the group of study subjects which will undergo control (sham) rehabilitation procedures (in addition to all their regularly scheduled treatments and interventions).

INTERVENTIONS:
Behavioral: Study-specific rehabilitation (SSR) procedures — Study-specific rehabilitation procedures will systematically manipulated the spatial or temporal synchrony (or coordination) of visual vs. haptic inputs that the subjects receive.
  Other Names: Study-related rehabilitation procedures
  Groups: Treatment Group

SUMMARY:
This study will help develop new methods of rehabilitating Veterans with vision loss due to Age-related macular degeneration.

DETAILED DESCRIPTION:
The purpose of this research study is to develop new and improved methods of helping vision-impaired Veterans see better by using hands as "seeing eyes". This study will focus on Veterans with a common form of eye disease called age-related macular degeneration that affects older individuals.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a Veteran.
2. The subject is 50 years of age.
3. The subject has best-corrected visual acuity (BCVA) of 20/40 or worse in each eye, as determined by the standard CNVAMC optometric tests.
4. The subject has visual field deficit of 10O in either eye as determined by the Octopus 900 perimetry (Haag-Streit Diagnostics, Haag-Streit USA, Mason, OH) administered by CNVAMC. (When the deficit/s are binocular, they do not necessarily have to be in binocularly corresponding positions.)
5. The subject has received a formal clinical diagnosis of age-related macular degeneration (AMD) in one or both eyes (binocular AMD does not necessarily have to be in binocularly corresponding positions)7,8,56.
6. The subject has visual deficit in either eye (wavy lines and/or missing/darkened areas on the grid) determined by the standard Amsler Grid Test7,8,56.
7. The subject has not yet started any rehabilitative treatment for AMD-related vision loss.
8. Both eyes of the subject are otherwise age-appropriately stable, and neither eye has any other visual defects, as determined by the standard CNVAMC ophthalmological examination.
9. The subject must be able to understand the nature and individual consequences of the study.
10. The subject must be able to provide signed and dated informed consent before start of any participation in the study procedures.
11. Women with childbearing potential must test negative for pregnancy using a standard urine test prior to participating in each functional magnetic resonance imaging (fMRI) procedure. (This exclusion criterion is mandated by the Augusta University Institutional Review Board [AU IRB], which also serves as the IRB of record of the CNVAMC. It is intended as an extra precautionary measure to help ensure the health and safety of this vulnerable population. The proposed study will comply with this requirement.)

Exclusion Criteria:

1. According to the patient's VA clinical records, the patient has one or more clinically diagnosed neurological disorder.
2. According to the patient's VA clinical records, the patient has one or more clinically diagnosed cognitive deficits.
3. According to the patient's VA clinical records, the patient has been clinically diagnosed with a psychiatric disorder that would make it unduly uncomfortable or otherwise clinically inadvisable for the subject to participate in the study.
4. According to the patient's VA clinical records, according to the patient, or both, the patient has motor disorder/s that would make it unduly uncomfortable or otherwise clinically inadvisable for the subject to participate in the study.
5. According to the patient's VA clinical records, according to the patient, or both, the patient has an MR-incompatible implant and/or another condition (e.g., claustrophobia) that would make it inadvisable for the subject to participate in MR imaging or any other study procedure.
6. The patient does not understand the informed consent information and/or the standard study instructions in spoken or written English, and/or is unable to follow study instructions. [The purpose of this exclusion criterion, required by the AU IRB, is to help ensure that the subjects adequately understand all the information relevant to providing informed consent, as well as the study instructions.]
7. Inability to give informed consent to participate in the study.
8. Pregnancy, as determined by a standard urine test for pregnancy.
9. Participation in other study/studies including an investigational drug or device during the present study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with vision loss caused by age-related macular degeneratioin
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of object recognition | 6-10 weeks
  This outcome will be measured as the accuracy (% correct) with which the study subjects recognize the text objects before, during and after their participation in the study procedures.
Response of brain regions of interest (ROI) as reflected in the BOLD (blood oxygenation level-dependent) response | 6-10 weeks
  This outcome will be measured as changes (if any) of the BOLD responses of brain ROIs before, during and after their participation in the study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hegde, PhD, Principal Investigator — Charlie Norwood VA Medical Center, Augusta, GA
Locations (1):
- Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No